CLINICAL TRIAL: NCT05013632
Title: COVID-19 International Drug Pregnancy Registry (COVID-PR)
Brief Title: COVID-19 International Drug Pregnancy Registry
Acronym: COVID-PR
Status: Recruiting | Type: Observational
Sponsor: Pregistry (Industry)
Responsible Party: Sponsor
Other Study IDs: PR005
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Antiviral Agents; remdesivir; molnupiravir; Antibodies, Monoclonal; casirivimab and imdevimab drug combination; casirivimab; imdevimab; sotrovimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Exposed pregnant women: Pregnant or recently pregnant women 18 years of age and older treated with monoclonal antibodies or antiviral drugs indicated for mild, moderate, or severe COVID-19 at any time during pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP.
  Interventions: Drug: Antiviral Agents; Drug: Monoclonal antibody
- Active comparator pregnant women: Pregnant women treated with another therapy for mild, moderate, or severe COVID-19
- Unexposed pregnant women: Pregnant women hospitalized but not treated with a medication specifically indicated for the treatment of mild, moderate, or severe COVID-19

INTERVENTIONS:
Drug: Antiviral Agents — Antiviral medications indicated for the treatment of mild to severe COVID-19
  Other Names: Veklury (remdesivir); Lagevrio (molnupiravir)
  Groups: Exposed pregnant women
Drug: Monoclonal antibody — Monoclonal antibodies indicated for the treatment of mild to severe COVID-19
  Other Names: REGEN-COV (casirivimab/imdevimab); Xevudy (sotrovimab)
  Groups: Exposed pregnant women

SUMMARY:
The objective of the COVID-19 International Drug Pregnancy Registry (COVID-PR) is to evaluate obstetric, neonatal, and infant outcomes among women treated with monoclonal antibodies or antiviral drugs indicated for mild, moderate, or severe COVID-19 from the first day of the last menstrual period (LMP) to end of pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP.

DETAILED DESCRIPTION:
Rationale and background: Pharmaceutical companies, academic centers, and other organizations globally are developing monoclonal antibodies and antiviral drugs to treat COVID-19. Pregnant women will be treated with these medications which, for the most part, lack scientific evidence regarding safety for the mother and the developing offspring.

Objective: To estimate the effect that monoclonal antibodies and antiviral drugs indicated for mild, moderate, or severe COVID-19 have on obstetric, neonatal, and infant outcomes.

Endpoints: Risk of obstetric outcomes (spontaneous abortion, intrauterine growth restriction, gestational diabetes, gestational hypertension, postpartum hemorrhage, Caesarean delivery), neonatal outcomes (major congenital malformations, low birth weight, small for gestational age, neonatal infections, stillbirth, neonatal death, preterm birth), and infant outcomes until 12 months of age (developmental milestones [motor, cognitive, language, social-emotional, and mental health skills], height, weight, failure to thrive).

Study design: The COVID-PR is an international, non-interventional, post-marketing cohort study designed to collect safety data among pregnant and recently pregnant women treated with monoclonal antibodies or antiviral drugs for mild, moderate, or severe COVID-19 from the first day of the last menstrual period (LMP) to end of pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP. Follow-up continues until the infant's first year of age.

Population: The study population includes pregnant or recently pregnant women 18 years of age and older treated with monoclonal antibodies or antiviral drugs indicated for mild, moderate, or severe COVID-19 at any time during pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP. Registration and participation via website especially developed for the COVID-PR are voluntary.

Eligible women can enroll at any time during pregnancy and up to 30 days after the end of pregnancy. Follow-up continues until the infant's first year of age.

Exposure: Women are considered exposed if they received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 at any time during pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP. The reference groups include pregnant women treated with another therapy for mild, moderate, or severe COVID-19 (active comparator) and pregnant women who were hospitalized for COVID-19 during pregnancy but were not treated with a medication specifically indicated for mild, moderate, or severe COVID-19 (unexposed comparator). The exposed and comparators are matched based on calendar time, country of residence, gestational week of COVID-19 infection (± 2 weeks), and severity of COVID-19.

Data collection: For women who enroll during pregnancy, the pregnancy information is collected at enrollment, monthly, and at the end of pregnancy. For women who enroll within 30 days after the end of pregnancy, the pregnancy and birth information (if there was a live birth) is collected at enrollment. Subsequently, data on liveborn infants are collected every three months until the infant's 12 months of age. Information is obtained directly from the participant. Detailed information is collected on COVID-19 symptoms, severity markers, and treatments. Additionally, a COVID-PR Clinical Research Associate calls the mother within 90 days after birth to answer any questions she may have about the registry and to request any missing information. The COVID-PR collects data on potential confounding factors (such as maternal sociodemographic characteristics, behaviors, reproductive history, use of assisted reproductive techniques, pre-pregnancy history of COVID-19 and test results, chronic conditions, use of medications, and measures of healthcare utilization) and detailed information associated with the obstetric, neonatal, and infant outcomes. In addition to self-reported information, the web-based data collection system requests medical records. Participants are asked to redact their personal identifiers, take photos of the label, container, or carton of the medication (if available), medical records from the hospital discharge, pediatric reports, and any other health care records they consider relevant and then upload them into the web-based data collection system. These records will be used to validate maternally reported diagnoses and to allow for potential future adjudication of outcomes. Given the international nature of the COVID-PR, the questionnaires are available in the languages spoken where it is conducted. Likewise, the phone call is conducted in the language spoken by the mother. Participant confidentiality and anonymity are strictly upheld.

Analysis: Exposure to medications indicated for mild, moderate, or severe COVID-19 during specific etiologically relevant periods will be considered when estimating the risk for each outcome (e.g., first trimester for miscarriages and malformations). Relative risks and their 95% confidence interval (CI) will be presented unadjusted and adjusted using propensity scores (PS) to account for imbalances in disease severity, comorbidities, and other characteristics between the exposed and the reference groups.

Study size: Monoclonal antibodies and antiviral drugs indicated for mild, moderate, or severe COVID-19 will be analyzed separately by brand. Efforts will be made to collect at least 100 pregnancies treated with each monoclonal antibody or antiviral drug during the first trimester and at least 100 exposed thereafter during pregnancy. For each exposed pregnancy, one pregnancy treated with another therapy for mild, moderate, or severe COVID-19 (active comparator) and one pregnancy with COVID-19 not treated with a medication specifically indicated for the treatment of mild to severe COVID-19 (unexposed comparator) will be matched based on calendar time, country of residence, gestational week of COVID-19 infection (± 2 weeks), and severity of COVID-19.

Milestones: The total duration of the study will be 5 years. Obstetric, neonatal, and infant outcomes will be assessed on an ongoing basis as data become available. The first two years will include, primarily, enrollment of pregnancies; the third and fourth years will involve follow-up of pregnancies and newborns; and, the final year, will be for data analyses and publications. Semi-annual and annual interim reports summarizing cumulative results on key outcomes will be submitted to the Scientific Advisory Committee (SAC) and to financial contributor pharmaceutical companies for their review and feedback every year of the study. A final report will be prepared at the end of the study.

Governance: The COVID-PR is conducted by Pregistry and includes an internal Safety Management Team (SMT) of experienced pharmacovigilance professionals and a dysmorphologist that meet regularly to review individual cases and safety signals. Additionally, the COVID-PR is in consultation with experts from relevant fields, such as maternal-fetal medicine, infectious diseases, epidemiology, and biostatistics from academic institutions and private practice. These individuals constitute the SAC and provide an independent review of the COVID-PR data.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or recently pregnant (up to 30 days after the end of pregnancy) at time of enrollment
* Age ≥18 years at time of enrollment
* With mild to severe COVID-19 during pregnancy
* Either

  * Treated for COVID-19 with at least one of the medications included in Table 1 during pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP or
  * Hospitalized and did not receive any pharmacological treatment specifically indicated for mild, moderate, or severe COVID-19 during pregnancy
* Resident of a country where a Central Institutional Review Board (IRB) or Ethics Committee provided approval to conduct the study or clearance that approval is not required to conduct the study
* Signed the informed consent form and submitted the baseline module "COVID-19 Medications During This Pregnancy"

Exclusion Criteria:

● <18 years of age

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: The exposed study population consists of pregnant or recently pregnant women 18 years of age and older treated with at least one dose of a monoclonal antibody or antiviral drug indicated for COVID-19 from first day of the LMP to end of pregnancy. For monoclonal antibodies, the exposure period also includes 90 days prior to the first day of the LMP. The reference groups include pregnant women not exposed to monoclonal antibodies or antiviral drugs and treated with another therapy for mild, moderate, or severe COVID-19 (active comparator) and women who experienced COVID-19 during pregnancy and were hospitalized but were not treated with a medication specifically indicated for mild, moderate, or severe COVID-19 (unexposed comparator), matched by calendar time, country of residence, gestational timing at the time of COVID-19 infection (± 2 weeks), and severity of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Obstetric outcomes | 1 year
  Number of pregnant women who received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 and number of pregnant women in the reference cohorts who experience spontaneous abortion, intrauterine growth restriction, gestational diabetes, gestational hypertension, postpartum hemorrhage, Caesarean delivery.
Neonatal outcomes | 1 year
  Number of newborns of women who received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 and number of newborns of pregnant women in the reference cohorts who experience major congenital malformations, low birth weight, small for gestational age, neonatal infections, stillbirth, neonatal death, preterm birth.
Infant weight | 1 year
  Change in weight from birth to 3, 6, 9, and 12 months of age among newborns of women who received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 and among newborns of pregnant women in the reference cohorts.
Infant developmental milestones | 1 year
  Change in developmental milestones from baseline at 6, 9, and 12 months based on the tool Caregiver Reported Early Development Instruments among the offspring of women who received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 and among the offspring of pregnant women in the reference cohorts.
Infant height | 1 year
  Change in length from birth to 3, 6, 9, and 12 months of age among newborns of women who received at least one dose of a monoclonal antibody or antiviral drug indicated for the treatment of mild, moderate, or severe COVID-19 and among newborns of pregnant women in the reference cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Renz, MD, Principal Investigator — Pregistry
Locations (1):
- Pregistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wyszynski DF, Papageorghiou AT, Renz C, Metz TD, Hernandez-Diaz S. The COVID-19 International Drug Pregnancy Registry (COVID-PR): Protocol Considerations. Drug Saf. 2024 Mar;47(3):195-204. doi: 10.1007/s40264-023-01377-2. Epub 2023 Nov 16. PMID 37973784
- See also: COVID-19 International Drug Pregnancy Registry (COVID-PR) — https://covid-pr.pregistry.com